CLINICAL TRIAL: NCT05633316
Title: Paired Non Inferiority Study Comparing Overture's Intracytoplasmic Sperm Injection Automated (ICSIA) System to the Standard Manual ICSI Process
Brief Title: Automated Intracytoplasmic Sperm Injection (ICSIA)
Acronym: ICSIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Overture Life (Industry)
Collaborators: New Hope Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09-21-2021_V1.0
Record Dates: First submitted 2022-10-31; First posted 2022-12-01 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: After the oocyte retrieval or thawing of donor oocytes, oocytes will be randomly assigned into equal groups: test and control. Test group oocytes will undergo ICSI via ICSIA (the investigational device), and control group oocytes will undergo manual ICSI as is routinely performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- ICSIA (Experimental): Intracytoplasmic sperm injection will be performed using the automated system named ICSIA (investigational device)
  Interventions: Device: Investigational device named ICSIA
- Control (Experimental): In this control group oocytes will undergo manual ICSI as is routinely performed.
  Interventions: Device: Manual ICSI

INTERVENTIONS:
Device: Investigational device named ICSIA — Oocytes will undergo intracytoplasmic sperm injection using the ICSIA (the investigational) device.
  Arms: ICSIA
Device: Manual ICSI — Oocytes will undergo intracytoplasmic sperm injection using the ICSI manual protocol
  Arms: Control

SUMMARY:
The purpose of this research study is to evaluate Overture's automated Intracytoplasmic Sperm Injection (ICSIA) System. ICSIA is an investigational medical device that automates injection of sperm into eggs. This study will evaluate survival and fertilization rates of oocytes handled via ICSIA and compare to survival and fertilization rates of oocytes which are manually injected with sperm.

DETAILED DESCRIPTION:
Today Intracytoplasmic Sperm Injection (ICSI) is performed manually; a highly skilled technician manually injects a single sperm cell into an oocyte using a set of microinjectors. Success of ICSI is contingent on operator skills and has a direct impact on the number of fertilized oocytes available and cumulative pregnancy rates. Automation of the ICSI technique may help improve consistency and efficiency of the process, as well as improve reproducibility across operators. Overture has developed the ICSI system to automate these critical processes, named ICSIA.

ICSIA is composed of the same devices and consumables used for manual ICSI, but these devices have been integrated using a software interface with artificial intelligence to identify oocytes and allow for proper puncture of the oocyte and injection of the sperm without human intervention. The information from this study will be used by the study Sponsor, Overture Life, Inc, to help future development of the System and for submission of data to the United States Food and Drug Administration (FDA).

During the study, patients will undergo a conventional IVF cycle, or donor IVF cycle. After the oocyte retrieval or thawing of donor oocytes, the oocytes will be placed into equal groups: test and control. Test group oocytes will undergo ICSI via ICSIA (the investigational device), and control group oocytes will undergo manual ICSI as is routinely performed. The oocytes will be immediately evaluated for survival and fertilization rates and remain separate for the duration of the study. ICSIA has been extensively tested in hamster and mice oocytes, and fertilization/survival rates after ICSIA have been between 89%-96%.

After ICSI, conventional IVF processes will be followed and fertilized oocytes cultured up to blastocyst stage. Blastocysts will be biopsied for preimplantation genetic testing for aneuploidy (PGT-A) which assesses the embryo's chromosomes. All biopsied blastocysts will be frozen, and frozen embryo transfers (FET) scheduled after genetic results have been received. Embryo freezing and thaw will be performed manually. Selection of the embryo for transfer (whether test or control) will be at random.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women undergoing IVF treatment with ICSI

Exclusion Criteria:

* Severe male factor infertility

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Infertile women undergoing IVF treatment
Enrollment: 10 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Survival rates | Between 0 hours and 2 hours post-ICSI
  It refers to the integrity of the oocytes after sperm injection out of the total number of oocytes injected.
Fertilization rates | Between 16 hours and 20 hours post-ICSI
  It refers to the number of oocytes that show to be correctly fertilized showing two pronuclei and a second polar body out of the total number of oocytes injected.

SECONDARY OUTCOMES:
Blastocyst rates | Between 120 hours and 168 hours post-ICSI
  Refers to the number of fertilized embryos that develop into a good quality blastocyst after 5-7 days of in vitro culture
Euploidy rates | 1 month after biopsy
  Refers to the number of blastocysts that are biopsied that are diagnosed as euploid
Clinical pregnancy rates | 6 weeks after embryo transfer
  Refers to the number of patients that are replaced with an embryo and result pregnant with fetal heartbeat out of the total patients that are transferred.

CONTACTS AND LOCATIONS:
Overall Officials: John Zhang, MD, Principal Investigator — New Hope Fertility Center
Locations (1):
- New Hope Fertility Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No